CLINICAL TRIAL: NCT00200109
Title: ONSTIM: Occipital Nerve Stimulation for the Treatment of Intractable Migraine.
Brief Title: Occipital Nerve Stimulation for the Treatment of Chronic Migraine Headache.
Acronym: ONSTIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1602
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Migraine Headache

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Other): See protocol
  Interventions: Device: Occipital Nerve Stimulation
- Group 2 (Other): See protocol
  Interventions: Device: Occipital Nerve Stimulation
- Group 3 (Other): See protocol
  Interventions: Device: Occipital Nerve Stimulation
- Group 4 (Other): See protocol
  Interventions: Device: Occipital Nerve Stimulation

INTERVENTIONS:
Device: Occipital Nerve Stimulation — Each group had a different plan

SUMMARY:
Background: Medically intractable chronic migraine (CM) is a disabling illness characterized by headache greater than 15 days per month.

Method: A multicenter, randomized, blinded, controlled feasibility study was conducted to obtain preliminary safety and efficacy data on occipital nerve stimulation (ONS) in CM. Eligible subjects received an occipital nerve block, and responsers were randomized to adjustable stimulation (AS), preset stimulation (PS) or medical management (MM) groups.

DETAILED DESCRIPTION:
The therapy under investigation involves a Medtronic neurostimulation device which delivers electrical impulses via insulated lead wires placed under the skin near the occipital nerves at the base of the head.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Migraine Headache by International Headache Society (IHS) criteria
* compliance with daily questionnaire
* headache that has not responded to at least two classes of headache medications
* stable headache medication regimen

Exclusion Criteria:

* previous surgical procedures to disrupt the nerves of the neck relating to the headache
* subjects who may require MRI or Diathermy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-05; Primary Completion 2008-06 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
A primary endpoint is not identified for this feasibility study. | No primary endpoint

SECONDARY OUTCOMES:
Secondary endpoints included: patient daily questionnaire, Migraine Disability Assessment (MIDAS), functional disability, SF-36, acute medication use and subject satisfaction surveys. | No secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Joel Saper, M.D., Principal Investigator — Michigan Head Pain and Neurological Institute, Ann Arbor, MI
Locations (9):
- United States (7):
  - Contact Medtronic for Exact Location, Scottsdale, Arizona
  - Contact Medtronic for Exact Locations, Oceanside, California
  - Contact Medtronic for Exact Locations, Denver, Colorado
  - Contact Medtronic for Exact Locations, Ann Arbor, Michigan
  - Contact Medtronic for Exact Locations, Detroit, Michigan
  - Contact Medtronic for Exact Locations, Oklahoma City, Oklahoma
  - Contact Medtronic for Exact Locations, Philadelphia, Pennsylvania
- Contact Medtronic for Exact Location, Calgary, Alberta, Canada
- Contact Medtronic for Exact Location, London, United Kingdom

REFERENCES:
- [Result] Saper JR, Dodick DW, Silberstein SD, McCarville S, Sun M, Goadsby PJ; ONSTIM Investigators. Occipital nerve stimulation for the treatment of intractable chronic migraine headache: ONSTIM feasibility study. Cephalalgia. 2011 Feb;31(3):271-85. doi: 10.1177/0333102410381142. Epub 2010 Sep 22. PMID 20861241